CLINICAL TRIAL: NCT06804226
Title: Advancing Discussions Using a Video-based Support Tool About End-of-life Care: the ADVISE Project
Brief Title: Advancing Discussions Using a Video-based Support Tool About End-of-life Care
Acronym: ADVISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Thaddeus J. Puzio, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HSC-MS-24-1256
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Traumatic Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video conversation aid (Experimental)
  Interventions: Behavioral: Video conversation aid
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Video conversation aid — A video conversation aid which provides information regarding life-sustaining care and encourages further goals of care discussions with a healthcare provider will be shown to patients or their surrogates (for those incapacitated and unable to make their own decisions) on admission or within 48 hours whenever feasible
  Arms: Video conversation aid
Behavioral: Usual Care — Participants and/or surrogates will participate in discussions surrounding life-sustaining care at healthcare provider discretion.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to evaluate the effectiveness and implementation considerations of a video aid to improve communication and patient-centered outcomes in older injured adults

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* admitted to any level of care following trauma

Exclusion Criteria:

* Prisoners
* Existing do not resuscitate (DNR)/do not intubate (DNI)
* Patients admitted while on hospice
* Patients not expected to survive over 24-48 hours

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who had a transition in code status from full code | at time of discharge (about 5 days after admission)
  Data will be reported categorically as number of participants who transitioned from full code to DNR/DNI, DNR, ok for intubation, or Comfort measures only

SECONDARY OUTCOMES:
Percentage of participants that recognize survival after Cardiopulmonary resuscitation (CPR) as less than 50 percent as assessed by a survey | at time of discharge (about 5 days after admission)
Number of participants that received information about life-sustaining care outcomes as assessed by a survey | at time of discharge (about 5 days after admission)
Number of participants that desire more information regarding life-sustaining care as assessed by a survey | at time of discharge (about 5 days after admission)
Number of participants that had hospital-free days | in the first 30 days after admission
Number of participants that had ICU-free days | at time of discharge (about 5 days after admission)
Discharge disposition | at time of discharge (about 5 days after admission)
  Data will be reported categorically as number of participants that were discharged to home, nursing facility, rehab facility, long term care hospital, hospice or number of participants that die
Number of participants that had ventilator-free days | at time of discharge (about 5 days after admission)
Decisional conflict score as assessed by the Decisional Conflict Scale | at time of discharge (about 5 days after admission)
  This is a 4 item questionnaire, each is scored as 0(no) or 1(yes), for a maximum score of 4, higher score indicating no decisional conflict
Number of interventional procedures | at time of discharge (about 5 days after admission)
  Procedures include tracheostomy, feeding tube placement, dialysis initiation

CONTACTS AND LOCATIONS:
Overall Officials: Thaddeus J Puzio, MD, MS, FACS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No